CLINICAL TRIAL: NCT02398695
Title: Oral Alkali Production and Caries Prevention in Children (Longitudinal Component)
Brief Title: Oral Alkali Production and Caries Prevention in Children (Longitudinal)
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 272-2012 SubStudy-N; K23DE023579 (NIH); IRB201600154 (Other: Univeristy of Florida)
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Dental Caries
Keywords: Plaque; Saliva; Caries
MeSH Terms: conditions — Dental Caries; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva and Plaque
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Caries Free: Participants who do not have caries (cavities) will have oral samples collected.
  Interventions: Other: Oral Samples
- Caries Active: Participants who do have caries (cavities) will have oral samples collected.
  Interventions: Other: Oral Samples

INTERVENTIONS:
Other: Oral Samples — Oral samples of saliva, dental plaque and DNA will be collected between the two groups.

SUMMARY:
The fact that dental caries remains a major public health problem mandates that oral-health researchers explore new strategies for assessment of caries risk, as well as for caries prevention and management. Dental caries occurs when acids produced by bacterial glycolysis of dietary carbohydrates causes demineralization of the tooth enamel. A major focus of caries research has been on identifying and characterizing acid-generating bacteria and the mechanisms of acid resistance. The purpose of this study is to investigate over time the relationship between alkali production and caries.

DETAILED DESCRIPTION:
This study will require a total of 6 study visits over a 2 to 3 year period. The first study visit will last about one hour. At this study visit, parent-administered questionnaires will be used to collect information on the following: (a) the participant's demographic background (age, gender, and race), (b) socio-economic status (parents' income and housing condition), (c) participant's oral health practice (feeding histories, diet habits, oral hygiene measures, and dental attendance), and (d) systemic diseases. During the study visit, the participant's complete medical and dental history will be obtained and reviewed, and a dental exam will be performed in order to determine participants' caries status, and intraoral pictures may be taken of participants' teeth. At this visit and remaining visits participants will not be allowed to brush or clean teeth using any type of oral hygiene procedures for 8 hours prior to the visit. Saliva and plaque (the solf white-yellowish material on the tooth surface) will be collected at each visit. The Investigator will use a small probe to measure the pH of the dental plaque that builds up on the teeth. The participant will be asked to dip one finger into a glass containing a buffer solution and the probe will be placed on the teeth from which plaque will be taken. Plaque samples will be collected by gently scrapping the tooth using a sterile instrument. If the participant does not have enough plaque samples, they will be asked to return on the following day.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to 7 years

Exclusion Criteria:

* Treated with antibiotics within the past 3 months
* taking any medication at the time of the study
* uses orthodontic appliance, and
* has performed oral hygiene procedures in the past 8 hour prior to the collection appointment.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will consist of unrelated children aged between 2 and 5 years with different levels of caries experience.
Sampling Method: Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2012-10; Primary Completion 2015-08-27 (Actual); Study Completion 2015-08-27 (Actual)

PRIMARY OUTCOMES:
Levels of the arginine deiminase system (ADS) in oral samples of healthy and caries-active subjects change from baseline to month 6. | Changes from baseline to month 6
  Saliva and dental plaque will be collected during the study visit. The amount of ammonia produced via the ADS by oral bacteria present in the collected oral samples will be measured using a standardized protocol.
Levels of the arginine deiminase system (ADS) in oral samples of healthy and caries-active subjects change from baseline to month 6 to month 12. | Changes from baseline to month 6 to month 12
  Saliva and dental plaque will be collected during the study visit. The amount of ammonia produced via the ADS by oral bacteria present in the collected oral samples will be measured using a standardized protocol.
Levels of the arginine deiminase system (ADS) in oral samples of healthy and caries-active subjects change from baseline to month 6 to month 12 to month 18. | Changes from baseline to month 6 to month 12 to month 18
  Saliva and dental plaque will be collected during the study visit. The amount of ammonia produced via the ADS by oral bacteria present in the collected oral samples will be measured using a standardized protocol.
Levels of the arginine deiminase system (ADS) in oral samples of healthy and caries-active subjects change from baseline to month 6 to month 12 to month 18 to month 24. | Changes from baseline to month 6 to month 12 to month 18 to month 24
  Saliva and dental plaque will be collected during the study visit. The amount of ammonia produced via the ADS by oral bacteria present in the collected oral samples will be measured using a standardized protocol.

SECONDARY OUTCOMES:
Bacteria collected from oral samples of healthy and caries-active subjects change from baseline to month 6. | Changes from baseline to month 6
  Saliva and dental plaque will be collected during the baseline study visit. These oral samples will be plated in specific medium for bacterial growth and isolation. The isolated bacteria will be identified by molecular and microbiological techniques to characterize their capacity to produce ammonia from arginine - ADS activity. Protocols will be used to determine the sensitivity of the ADS of the oral isolates to environmental oral factors.
Bacteria collected from oral samples of healthy and caries-active subjects change from baseline to month 6 to month 12. | Changes from baseline to month 6 to month 12
  Saliva and dental plaque will be collected during the baseline study visit. These oral samples will be plated in specific medium for bacterial growth and isolation. The isolated bacteria will be identified by molecular and microbiological techniques to characterize their capacity to produce ammonia from arginine - ADS activity. Protocols will be used to determine the sensitivity of the ADS of the oral isolates to environmental oral factors.
Bacteria collected from oral samples of healthy and caries-active subjects change from baseline to month 6 to month 12 to month 18. | Changes from baseline to month 6 to month 12 to month 18,
  Saliva and dental plaque will be collected during the baseline study visit. These oral samples will be plated in specific medium for bacterial growth and isolation. The isolated bacteria will be identified by molecular and microbiological techniques to characterize their capacity to produce ammonia from arginine - ADS activity. Protocols will be used to determine the sensitivity of the ADS of the oral isolates to environmental oral factors.
Bacteria collected from oral samples of healthy and caries-active subjects change from baseline to month 6 to month 12 to month 18 to month 24. | Changes from baseline to month 6 to month 12 to month 18 to month 24.
  Saliva and dental plaque will be collected during the baseline study visit. These oral samples will be plated in specific medium for bacterial growth and isolation. The isolated bacteria will be identified by molecular and microbiological techniques to characterize their capacity to produce ammonia from arginine - ADS activity. Protocols will be used to determine the sensitivity of the ADS of the oral isolates to environmental oral factors.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelle Nascimento, DDS, MS, PhD, Principal Investigator — University of Florida
Locations (1):
- Dental Clinical Research Unit, University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Nascimento MM, Liu Y, Kalra R, Perry S, Adewumi A, Xu X, Primosch RE, Burne RA. Oral arginine metabolism may decrease the risk for dental caries in children. J Dent Res. 2013 Jul;92(7):604-8. doi: 10.1177/0022034513487907. Epub 2013 May 2. PMID 23640952